CLINICAL TRIAL: NCT05165966
Title: A Randomized, Double-Blinded Clinical Trial to Evaluate the Immunogenicity Using Additional Dose of Medium-dosage or High-dosage COVID-19 Vaccine (Vero Cell), Inactivated in Populations Who Have Completed Primary Immunization 5-9 Months
Brief Title: Safety and Immunogenicity Study of Booster Vaccination in Different Doses of COVID-19 Vaccine (Vero Cell),Inactivated for Prevention of COVID-19
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac Life Sciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO-nCOV-4010
Record Dates: First submitted 2021-12-20; First posted 2021-12-21 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2021-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — sinovac COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group-High-dosage of COVID-19 vaccine (Vero cell), Inactivated (Experimental): 170 participants will receive one dose of booster vaccination with high-dosage of COVID-19 vaccine (Vero cell), Inactivated.
  Interventions: Biological: High-dosage of COVID-19 vaccine (Vero cell), Inactivated
- Experimental Group-Medium-dosage of COVID-19 vaccine (Vero cell), Inactivated (Experimental): 170 participants will receive one dose of booster vaccination with medium-dosage of COVID-19 vaccine (Vero cell), Inactivated.
  Interventions: Biological: Medium-dose COVID-19 Vaccine(Vero Cell),Inactivated

INTERVENTIONS:
Biological: High-dosage of COVID-19 vaccine (Vero cell), Inactivated — High-dose COVID-19 Vaccine(Vero Cell),Inactivated:1200SU inactivated SARS-CoV-2 virus in 0.5 mL of aluminium hydroxide solution per injection
  Other Names: High-dose CoronaVac®
  Arms: Experimental Group-High-dosage of COVID-19 vaccine (Vero cell), Inactivated
Biological: Medium-dose COVID-19 Vaccine(Vero Cell),Inactivated — Medium-dose COVID-19 Vaccine(Vero Cell),Inactivated: 600SU inactivated SARS-CoV-2 virus in 0.5 mL of aluminium hydroxide solution per injection
  Other Names: Medium-dose CoronaVac®
  Arms: Experimental Group-Medium-dosage of COVID-19 vaccine (Vero cell), Inactivated

SUMMARY:
This is a randomized, double-blinded, phase Ⅳ clinical trial of COVID-19 vaccine (Vero cell), Inactivated manufactured by Sinovac Life Sciences Co. , Ltd. The purpose of this study is to evaluate the safety and immunogenicity of booster vaccination using high-dosage or medium-dosage of COVID-19 vaccine (Vero cell), Inactivated in populations who have completed primary immunization 5-9 months

DETAILED DESCRIPTION:
This study a randomized, double-blinded, phase Ⅳ clinical trial of COVID-19 vaccine (Vero cell), Inactivated.The purpose of this study is to evaluate the safety and immunogenicity of booster vaccination using high-dosage or medium-dosage of COVID-19 vaccine (Vero cell), Inactivated in populations who have completed primary immunization 5-9 months.A total of 340 subjects who have completed primary immunization using two-dose Coronavac® 5-9 months were be enrolled.All of subjects were be randomly divided into two groups in a 1:1 ratio to receive high-dosage or medium-dosage of COVID-19 vaccine (Vero cell), Inactivated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants aged 18 years and above;
* Proven legal identity;
* The subjects can understand and voluntarily sign the informed consent form and be willing to complete the study in accordance with the study plan;
* Have received two doses of inactivated COVID-19 vaccine (CoronaVac®) manufactured by Sinovac Research & Development Co., Ltd and that is currently 5-9 months after the second dose.

Exclusion Criteria:

* History of SARS-CoV-2 infection(laboratory confirmed);
* Have received three and more doses of inactivated COVID-19 vaccine;
* Known allergy to vaccines or vaccine ingredients, and serious adverse reactions to vaccines, such as urticaria, dyspnea, angioneurotic edema;
* Autoimmune disease such as systemic lupus erythematosus or immunodeficiency / immunosuppression such as AIDS, post-transplant;
* Severe chronic diseases, severe cardiovascular diseases, hypertension and diabetes that cannot be controlled by drugs, liver or kidney diseases, malignant tumors, etc;
* Severe neurological disease (epilepsy, convulsions or convulsions) or mental illness;
* Diagnosed abnormal blood coagulation function (eg, lack of blood coagulation factors, blood coagulopathy, abnormal platelets) or obvious bruising or blood coagulation;
* Immunosuppressive therapy, cytotoxic therapy, inhaled corticosteroids(excluding allergic rhinitis corticosteroid spray therapy, acute noncomplicated dermatitis superficial corticosteroid therapy) in the past 6 months;
* History of alcohol or drug abuse;
* Receipt of blood products within in the past 3 months;
* Receipt of other investigational drugs in the past 30 days;
* Receipt of attenuated live vaccines in the past 14 days;
* Acute diseases or acute exacerbation of chronic diseases within 7 days prior to booster vaccination;
* Axillary temperature >37.0°C;
* Participated in other clinical trials prior to enrollment and during the followup period, or planned to participate in other clinical trials during the clinical trial period;
* According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Immunogenicity index-GMT of neutralizing antibodies(CZ02 strain) | 14 days after the booster dose vaccination
  GMT of neutralizing antibodies(CZ02 strain) 14 days after the booster dose vaccination

SECONDARY OUTCOMES:
Immunogenicity index-Seropositivity rate of neutralizing antibodies(CZ02 strain) | 14 days after the booster dose vaccination
  Seropositivity rate of neutralizing antibodies(CZ02 strain) 14 days after the booster dose vaccination

OTHER OUTCOMES:
Immunogenicity index-GMI of neutralizing antibodies(CZ02 strain) | 14 days after the booster dose vaccination
  GMI of neutralizing antibodies(CZ02 strain) 14 days after the booster dose vaccination
Immunogenicity index-seroconversion rate of neutralizing antibodies(CZ02 strain) | 14 days after the booster dose vaccination
  The seroconversion rate of neutralizing antibodies(CZ02 strain) 14 days after the booster dose vaccination
Immunogenicity index-GMT of neutralizing antibodies(CZ02 strain) | 7 days after the booster dose vaccination
  GMT of neutralizing antibodies(CZ02 strain) 7 days after the booster dose vaccination
Immunogenicity index-Seropositivity rate of neutralizing antibodies(CZ02 strain) | 7 days after the booster dose vaccination
  Seropositivity rate of neutralizing antibodies(CZ02 strain) 7 days after the booster dose vaccination
Immunogenicity index-GMI of neutralizing antibodies(CZ02 strain) | 7 days after the booster dose vaccination
  GMI of neutralizing antibodies(CZ02 strain)7 days after the booster dose vaccination
Immunogenicity index-seroconversion rate of neutralizing antibodies(CZ02 strain) | 7 days after the booster dose vaccination
  The seroconversion rate of neutralizing antibodies(CZ02 strain) 7 days after the booster dose vaccination
Immunogenicity index-GMT of neutralizing antibodies(CZ02 strain) | 28 days after the booster dose vaccination
  GMT of neutralizing antibodies(CZ02 strain) 28 days after the booster dose vaccination
Immunogenicity index-Seropositivity rate of neutralizing antibodies(CZ02 strain) | 28 days after the booster dose vaccination
  Seropositivity rate of neutralizing antibodies(CZ02 strain) 28 days after the booster dose vaccination
Immunogenicity index-GMI of neutralizing antibodies(CZ02 strain) | 28 days after the booster dose vaccination
  GMI of neutralizing antibodies(CZ02 strain)28 days after the booster dose vaccination
Immunogenicity index-seroconversion rate of neutralizing antibodies(CZ02 strain) | 28 days after the booster dose vaccination
  The seroconversion rate of neutralizing antibodies(CZ02 strain) 28 days after the booster dose vaccination
Immunogenicity index-GMT of neutralizing antibodies(CZ02 strain) | 3 months after the booster dose vaccination
  GMT of neutralizing antibodies(CZ02 strain) 3 months after the booster dose vaccination
Immunogenicity index-seroconversion rate of neutralizing antibodies(CZ02 strain) | 3 months after the booster dose vaccination
  The seroconversion rate of neutralizing antibodies(CZ02 strain)3 months after the booster dose vaccination
Immunogenicity index-GMT of neutralizing antibodies(CZ02 strain) | 6 months after the booster dose vaccination
  GMT of neutralizing antibodies(CZ02 strain) 6 months after the booster dose vaccination
Immunogenicity index-GMT of neutralizing antibodies(Delta strain) | 14 days after the booster dose vaccination
  GMT of neutralizing antibodies(Delta strain) 14 days after the booster dose vaccination
Immunogenicity index-Seropositivity rate of neutralizing antibodies(Delta strain) | 14 days after the booster dose vaccination
  Seropositivity rate of neutralizing antibodies (Delta strain) 14 days after the booster dose vaccination
Immunogenicity index-GMI of neutralizing antibodies(Delta strain) | 14 days after the booster dose vaccination
  GMI of neutralizing antibodies(Delta strain) 14 days after the booster dose vaccination
Immunogenicity index-seroconversion rate of neutralizing antibodies(Delta strain) | 14 days after the booster dose vaccination
  The seroconversion rate of neutralizing antibodies (Delta strain) 14 days after the booster dose vaccination
Immunogenicity index-GMT of neutralizing antibodies(Omicron Strain) | 14 days after the booster dose vaccination
  GMT of neutralizing antibodies(Omicron Strain) 14 days after the booster dose vaccination
Immunogenicity index-Seropositivity rate of neutralizing antibodies(Omicron Strain) | 14 days after the booster dose vaccination
  Seropositivity rate of neutralizing antibodies (Omicron Strain) 14 days after the booster dose vaccination
Immunogenicity index-GMI of neutralizing antibodies(Omicron Strain) | 14 days after the booster dose vaccination
  GMI of neutralizing antibodies(Omicron Strain) 14 days after the booster dose vaccination
Immunogenicity index-seroconversion rate of neutralizing antibodies(Omicron Strain) | 14 days after the booster dose vaccination
  The seroconversion rate of neutralizing antibodies (Omicron Strain) 14 days after the booster dose vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Yingmei Feng, Master, Principal Investigator — Beijing YouAn Hospital
Locations (1):
- Beijing Youan Hospital Capital Medical University, Beijing, Beijing Municipality, China